CLINICAL TRIAL: NCT01962168
Title: Palliation of Biliary Neoplasms With the Cook Evolution® Biliary Stent System
Brief Title: Evolution® Biliary Stent System Clinical Study
Status: Completed | Type: Observational
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: 12-009
Record Dates: First submitted 2013-10-09; First posted 2013-10-14 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Biliary Tract Neoplasms; Neoplasms; Gastrointestinal Diseases; Digestive System Diseases; Biliary Tract; Stents
Keywords: Biliary Tract Neoplasms; Neoplasms; Gastrointestinal Diseases; Digestive System Diseases; Biliary Tract; Stents
MeSH Terms: conditions — Biliary Tract Neoplasms; Neoplasms; Gastrointestinal Diseases; Digestive System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Evolution® Biliary Stent - Uncovered
  Interventions: Device: Evolution® Biliary Stent - Uncovered

INTERVENTIONS:
Device: Evolution® Biliary Stent - Uncovered — Commercially available device

SUMMARY:
The Evolution® Biliary Stent System Clinical Study is a clinical trial on a commercially available device to gather physician experience with the Cook Evolution® Biliary Stent System for the palliation of cancer in the biliary tree. Patients will be treated as per usual medical practices.

ELIGIBILITY:
Inclusion Criteria:

* Patient is considered a candidate for stent placement based on institutional guidelines and product IFU.

Exclusion Criteria:

* Patient is less than 18 years of age.
* Patient is unable or unwilling to provide written informed consent.
* Patient is unable or unwilling to comply with the follow-up schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Candidates for biliary stent placement based on institutional guidelines and product IFU.
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2013-12; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Freedom from symptomatic recurrent biliary obstruction requiring reintervention | 6 months

SECONDARY OUTCOMES:
Technical success | Immediately following completion of the stent placement procedure
  Technical success is defined as a stent successfully delivered and placed at its intended location at the end of the procedure.
Incidence of device-related adverse events | 6 months
Ease of use | Immediately following completion of the stent placement procedure
  Ease of use will be evaluated on a five point scale ranging from very easy to very difficult.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Lawrence, Principal Investigator — Summerville GI & Advanced Endoscopy
Locations (9):
- United States (8):
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - The Pancreas and Biliary Center of South Florida, Boca Raton, Florida
  - Borland-Groover Clinic, Jacksonville, Florida
  - Florida Hospital, Orlando, Florida
  - Northwest Community Hospital, Arlington Heights, Illinois
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - SUNY at Stony Brook Hospital, Stony Brook, New York
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
- Centre Hospitalier de l' Universite de Montreal (CHUM), Montreal, Quebec, Canada

REFERENCES:
- [Derived] Lawrence C, Nieto J, Parsons WG, Roy A, Guda NM, Steinberg SE, Hasan MK, Bucobo JC, Nagula S, Dey ND, Buscaglia JM; Study Investigators. A newly designed uncovered biliary stent for palliation of malignant obstruction: results of a prospective study. BMC Gastroenterol. 2020 Jun 10;20(1):184. doi: 10.1186/s12876-020-01325-9. PMID 32522161